CLINICAL TRIAL: NCT00714220
Title: Quantitative Measurement of Nutritional Substrate Utilization in Patients With ALS
Brief Title: Quantitative Measurement of Nutritional Substrate Utilization in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Type: Observational
Why Stopped: Lack of funding and support staff.
Sponsor: Drexel University College of Medicine (Other)
Collaborators: MDA/ALS Center of Hope (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Other Study IDs: Internal-16684
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases
Keywords: Amyotrophic Lateral Sclerosis; Gastric Motility; Autonomic Nervous System; Neurodegenerative Diseases; Movement Disorders; Substrate Utilization
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- ALS: Subjects having either definite or probable ALS by El Escorial Criteria.
- Neurological Control: Subjects having been diagnosed with a non-ALS neurological condition
- Healthy Control: Subjects in good health without any neurological conditions

SUMMARY:
The work of Nau et. al (Nau KL, Bromberg MB, Forshew DA, Katcha Vl. Individuals with amyotrophic lateral sclerosis are in caloric balance despite losses in mass. J Neurol Sci 1995;129 :47-49) showed that patients in the early stages of ALS initially increase their body fat. Another study showed that advanced ALS patients on mechanical ventilation were actually hypometabolic, supporting a hypothesis that ALS patients' daily oral intakes of calories fail to match their energy requirements, thus exacerbating their condition. This current study investigates and compares substrate utilization using a metabolic cart in controls and in ALS patients who are on and off ventilatory support to examine differences in substrate utilization between the two groups of ALS patients and the controls. (Substrate utilization is essentially the percentage of fats, carbohydrates, and protein utilized by the body.) The study will increase our understanding of the nutritional needs of ALS patients and improve our ability to provide the best possible nutrition in progressive illness.

DETAILED DESCRIPTION:
Study groups will include ALS patients with and without respiratory failure as judged by their FVC and use of either noninvasive or invasive ventilation along with normal controls. For all patients, nutritional status will be assessed by measurement of weight, and determination of Urinary Urea Nitrogen (via 24hr urinary sample), albumin and pre-albumin levels and questions regarding recent weight changes. In addition, for ALS patients, clinical data regarding the age of the patient, duration of disease, site of onset along with ALS-FRS (Amyotrophic Lateral Sclerosis Functional Rating Scale) and Pulmonary function testing will be collected. If these data are already available from chart as they are commonly performed during routine care, the data will be obtained from the patients chart.

5cc blood will be obtained for measurement of Serum albumin, pre-albumin and TNF-α. Antigenic TNF-α, bioactive TNF-α and receptors serum sTNF-RI and TNF-RII will be measured using the standard ELISA kits and cytolytic assays.

Respiratory Quotients (RQs) will be measured using a metabolic cart in both controls and ALS patients. First, the patient's VCO2 and VO2 will be measured - as the patient breaths into a mask connected to the machine.- RQ will be calculated using Lavoisier and Laplace's equation: RQ = VCO2/VO2.

This, however, is not an accurate representation because it considers only fats and carbohydrates as the sources for these gases. A corrected Non-Protein RQ (NPRQ) RQ will be calculated using a 24 hour urine sample and measuring the Urinary Urea Nitrogen (24hr UUN). This tells us the amount of protein oxidized per 24 hours. Then, applying the principle that one gram of urinary nitrogen represents the combustion of an amount of protein that requires 5.925L of oxygen and produces 4.75L of carbon dioxide, the amount of oxygen and carbon dioxide associated with protein metabolism will be calculated. This calculated VO2 and VCO2 will then be subtracted from the totals measured using the metabolic cart and the corrected Non-Protein RQ will be calculated.

The corrected respiratory quotient will then be used to calculate the amount of nutritional substrate utilization in the patient population using Table 7.2. Non-Protein Respiratory Quotient And The Relative Quantity Of Carbohydrate And Fat Oxidized And Energy Per Liter Of Oxygen (Appendix-I).v The amount (grams) of carbohydrate and fats utilized per each NPRQ will be recorded.

The protein catabolic rate (PCR) will also be calculated using the equation :

PCR=[24hr UUN(g) + 4] x 6.25 (g/day). The clinical information along with test results will be collected in a spreadsheet in which patients and controls are de-identified. This spreadsheet will be used for the analysis.

Primary endpoints are the analysis of nutritional substrate utilization with and without respiratory compromise. Secondary endpoints include the correlation of in the composition of substrate utilization between patients who use a ventilator and those who do not, those patients with and without a PEG Tube in each group, and correlation of substrate use with the stage of illness as judged by the ALSFRS score, weight changes and duration of disease.

This is a one time testing procedure, and the patient will not be asked to return back for another visit.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of definite or possible ALS by the El Escorial Criteria
* No previously known gastrointestinal problems

Exclusion Criteria:

* Patients or controls who have evidence of previous gastrointestinal disease
* Patients unable to give informed consent

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS clinic patients at MDA/ALS Center of Hope.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2006-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Indirect Calorimetry | 20 minute session
  Indirect calorimetry will be used to determine how many calories you are burning and how much of your total calories burned are fats.

CONTACTS AND LOCATIONS:
Locations (1):
- MDA/ALS Center of Hope, Philadelphia, Pennsylvania, United States